CLINICAL TRIAL: NCT00000172
Title: Placebo Controlled Evaluation of Galantamine in the Treatment of Alzheimer's Disease: Safety and Efficacy Under a Slow-Titration Regimen
Brief Title: Evaluation of Galantamine in the Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0009
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Cholinergic agents; Cholinergic agonists; Cholinesterase inhibitors
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine

SUMMARY:
Galantamine is an experimental drug being evaluated in the United States for the treatment of Alzheimer's disease. Results from previous clinical trials suggest that galantamine may improve cognitive performance in individuals with Alzheimer's disease. It is not a cure for Alzheimer's disease. Nerve cells in the brain responsible for memory and cognitive function communicate using a chemical called acetylcholine. Research has shown that deterioration of cells that produce acetylcholine in the brain affects thought processes. Galantamine is thought to work in two ways to increase the amount of acetylcholine available in the brain. It inhibits an enzyme that breaks down acetylcholine and it also stimulates the nicotinic receptors in the brain to release more acetylcholine.

DETAILED DESCRIPTION:
After a 1-month single-blind run in phase, 910 subjects will be titrated, over a period of up to 8 weeks, to target doses of either: 0 (placebo); 24 mg/day galantamine; 16 mg/day galantamine; or 8 mg/day galantamine, in a 2:2:2:1 randomization ratio. Double-blind treatment will continue for a total of 5 months. The change from baseline in ADAS-cog and CIVIC-plus scores at Month 5 will be the primary efficacy endpoints. Tolerability will be evaluated based on adverse event reports, laboratory values, ECG, and vital signs with particular focus on the adverse event rates in the slower titration schedule for 24 mg/day. Efficacy of 24 mg/day and 16 mg/day galantamine will be compared with that of placebo. Information on the dose response relationship of galantamine will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease
* Mini-Mental State Examination (MMSE) 10-22 and ADAS greater than or equal to 18
* Alzheimer's Disease Assessment Scale cognitive portion (ADAS-cog-11) score of at least 18
* Opportunity for Activities of Daily Living
* Caregiver
* Subjects who live with or have regular daily visits from a responsible caregiver (visit frequency: preferably daily but at least 5 days/week). This includes a friend or relative or paid personnel. The caregiver should be capable of assisting with the subject's medication, prepared to attend with the subject for assessments, and willing to provide information about the subject.

Exclusion Criteria:

* Conditions that could confound diagnosis
* Neurodegenerative disorders
* Acute cerebral trauma
* Psychiatric disease
* More than one infarct on CT/MRI scans
* History of alcohol or drug abuse
* Contradictions for a cholinominetic agent: seizures; ulcers; pulmonary conditions (including severe asthma); unstable angina; Afib; bradycardia less than 50; and AV block.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (55):
- United States (55):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - James L. Frey, M.D., Ltd., Scottsdale, Arizona
  - East Bay Neurology, Berkeley, California
  - University of Southern California, Los Angeles, California
  - N. County Neurology Assoc., Oceanside, California
  - University of California Irvine Medical Center, Orange, California
  - Pacific Research Network (PRN), San Diego, California
  - Affiliated Research Institute, San Diego, California
  - INC, San Diego, California
  - The Denver Center for Medical Research, Denver, Colorado
  - Geriatric and Adult Psychiatry, Hamden, Connecticut
  - Yale University, School of Medicine, New Haven, Connecticut
  - Ocala Neurodiagnostic Center, Ocala, Florida
  - Psychiatric Institute of Florida, Orlando, Florida
  - Neurological Research Institute of Sarasota, PA, Sarasota, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Chicago Center for Clinical Research, Chicago, Illinois
  - OSF Center for Senior Health, Peoria, Illinois
  - Indiana Alzheimer's University Clinic, Indianapolis, Indiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham Behavioral Neurology Group, Boston, Massachusetts
  - Boston Clinical Research Center, Wellesley Hills, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Michigan Medical P.C., Grand Rapids, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - St. Louis University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - University of Medicine and Dentistry of New Jersey, Piscataway, New Jersey
  - Neurology Group of Bergen County, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Medwise Center, West Long Branch, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - East End Neuropsychiatric Associates, Centereach, New York
  - St. John's Episcopal Hospital, Far Rockaway, New York
  - NYU Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Ohio State University, Columbus, Ohio
  - Clinical Pharmaceutical Trials, Tulsa, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Pacific NW Clinical Research Center, Portland, Oregon
  - Institute for Advanced Clinical Research, Elkins Park, Pennsylvania
  - Neuroscience Center of Westmoreland Neurology, Greensburg, Pennsylvania
  - Brown University, Pawtucket, Rhode Island
  - Alzheimer's Research and Clinical Programs, North Charleston, South Carolina
  - University of Texas, Dallas, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Memory Disorder Center of Vermont, Colchester, Vermont
  - Virginia Neuroscience Center, Alexandria, Virginia
  - Prince William Neuroscience Center, Manassas, Virginia
  - Seattle Clinical Research Center, Seattle, Washington
  - VAPS Health Care System, Seattle, Washington

REFERENCES:
- [Background] Lilienfeld S, Parys W. Galantamine: additional benefits to patients with Alzheimer's disease. Dement Geriatr Cogn Disord. 2000 Sep;11 Suppl 1:19-27. doi: 10.1159/000051228. PMID 10971048